CLINICAL TRIAL: NCT03489395
Title: A Pilot Study on Edoxaban for the Resolution of Left Atrial Thrombosis in Patients With Non-valvular Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raffaele De Caterina (Other)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor-Investigator, Raffaele De Caterina, Professor, G. d'Annunzio University
Organization: G. d'Annunzio University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDO-SP-01-2015; 2015-004847-37 (EudraCT Number)
Record Dates: First submitted 2018-03-15; First posted 2018-04-05 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Intervention Model Description: Non-controlled, open-label pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Edoxaban (Experimental): Used for Treatment. All patients will receive edoxaban 60 mg once a day, with open-label design, for 4 weeks. Edoxaban daily dose will be reduced to 30 mg/day in case of: body weight ≤60 kg, or concomitant therapy with verapamil/quinidine/dronedarone.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 60 mg once a day for 4 weeks. Edoxaban 30 mg/day in patients with body weight ≤60 kg, or with concomitant therapy with verapamil/quinidine/dronedarone.
  Other Names: Lixiana

SUMMARY:
Isolated reports have indicated that complete Left Atrial or Left Atrial Appendage thrombus resolution may be achieved also with use of oral Factor Xa inhibitors, which have demonstrated the same efficacy but a better safety profile compared to warfarin.

The aim of this open-label pilot study is to investigate the percentage of Left Atrial /Left Atrial Appendage thrombus resolution with edoxaban therapy in patients with non-valvular atrial fibrillation. The subordinated aim is the design a larger and longer study to compare edoxaban and warfarin in the same patient population.

With the exception of few case reports, there are no data in the same patient population referred to antithrombotic treatments other than vitamin K antagonists.

DETAILED DESCRIPTION:
This is a non-controlled, open-label, 4 weeks pilot study.

As the main goal of this exploratory study is the estimation of the magnitude of the Left Atrial /Left Atrial Appendage thrombus resolution with edoxaban, no control group with vitamin K antagonists has been considered, providing that, for the purpose of this study, the magnitude of the response of warfarin is satisfactory defined.

ELIGIBILITY:
Inclusion Criteria:

Patients with all the following criteria will be eligible for inclusion in the study protocol:

1. Signed written informed consent.
2. Males and females ≥ 18 years of age.
3. Female subjects must be post-menopausal (for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and, for those of childbearing potential, have a negative serum β-human chorionic gonadotropin pregnancy test at screening.
4. Atrial fibrillation (AF) must be documented by ECG evidence (e.g., 12-lead ECG, rhythm strip, Holter, pacemaker interrogation) within 30 days before enrolment.
5. Subjects with newly diagnosed atrial fibrillation are eligible provided that:

   * -there is evidence that the atrial fibrillation is non-valvular:
   * -there is ECG evidence on 2 occasions 24 hours apart demonstrating atrial fibrillation.
6. Left Atrial or Left Atrial Appendage thrombosis documented by trans-esophageal echocardiography (TEE)
7. Cardiac failure, Hypertension, Age (x2 ), Diabetes, Stroke (x 2) risk index-VASC score >1.

Exclusion Criteria:

Patients with all the following criteria will not be eligible for inclusion in the study protocol:

1. Hemodynamically significant mitral valve stenosis.
2. Prosthetic heart mechanical or biological valve (annuloplasty with or without prosthetic ring, commissurotomy and/or valvuloplasty are permitted).
3. Transient atrial fibrillation caused by a reversible disorder (e.g., thyrotoxicosis, pulmonary embolism, recent surgery or myocardial infarction).
4. Known presence of atrial myxoma.
5. Left ventricular thrombus.
6. Active endocarditis.
7. Active internal bleeding.
8. History of condition associated with increased bleeding risk including, but not limited to:

   * major surgical procedure or trauma within 30 days;
   * clinically significant gastrointestinal bleeding within 6 months;
   * previous intracranial, intraocular, spinal, atraumatic intra-articular bleeding;
   * chronic haemorrhagic disorder;
   * Any neoplasm, including intracranial neoplasm,
   * arteriovenous malformation or aneurysm.
9. Platelet count <90,000/μL at the screening visit.
10. Sustained uncontrolled hypertension: Systolic Blood Pressure ≥180 mmHg or Diastolic Blood Pressure ≥100 mmHg.
11. Severe, disabling stroke (modified Rankin score of 4 to 5, inclusive within 3 months or any stroke < 14 days).
12. Transient ischemic attack within 3 days.
13. Any oral anticoagulant therapy at the time of the baseline visit.
14. Treatment with:

    * aspirin >160 mg daily;
    * aspirin plus a thienopyridine within 5 days;
    * intravenous antiplatelets within 5 days;
    * fibrinolytics within 10 days.
15. Anticipated need for therapy with a non-steroidal anti-inflammatory drug in the next 4 weeks.
16. Treatment with a strong inducer of cytochrome P450 and P glycoprotein, such as ketoconazole, itraconazole, voriconazole, posaconazole, ritonavir, lopinavir, telaprevir, indinavir, conivaptan, clarithromycin or planned treatment during the study.
17. Other indication for anticoagulant therapy.
18. Hypersensitivity or intolerance to the study drug, including excipients.
19. Women of childbearing potential who do not want adopt a contraceptive method during the study period and the following 4 weeks.
20. Breast-feeding women during the study period and the following 4 weeks.
21. Anemia (hemoglobin <10 g/dL) at the screening visit.
22. Known significant liver disease (e.g., acute clinical hepatitis, chronic active hepatitis, cirrhosis), or Alanine aminotransferase or Aspartate aminotransferase >2 x Upper Level of Normal or total bilirubin >1.5 x Upper Level of Normal.
23. Patients with moderate or severe renal impairment (CrCL <50 mL/min) or patients with end stage renal disease (CrCL < 15 mL/min) or on dialysis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete thrombus resolution by TEE, evaluated with the following Probe angulations: 0°, 45°-to-60°, 90°. | 4 weeks
  Only a descriptive statistical analysis will be performed.

SECONDARY OUTCOMES:
Absolute variation of thrombus area by TEE evaluation (Probe angulations: 0°, 45-to-60°, 90°) | 4 weeks
  Only a descriptive statistical analysis will be performed.
Percent variation of thrombus area by TEE evaluation (Probe angulations: 0°, 45-to-60°, 90°) | 4 weeks
  Only a descriptive statistical analysis will be performed.
Time to electrical cardioversion (when applicable). | 4 weeks
  Only a descriptive statistical analysis will be performed.

OTHER OUTCOMES:
Safety analysis - Percentage of bleeding events (telephone assessment) | 4 weeks and 8 weeks
  Only a descriptive statistical analysis will be performed.
Safety analysis - Percentage of any stroke or peripheral embolism (telephone assessment) | 4 weeks and 8 weeks
  Only a descriptive statistical analysis will be performed.
Safety analysis - Percentage of any other safety related events (deaths, Serious Adverse Events and Adverse Events). | 4 weeks and 8 weeks
  Only a descriptive statistical analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele De Caterina, Principal Investigator — Università degli Studi G. d'Annunzio Chieti
Locations (8):
- Italy (8):
  - Ospedale Madonna del Soccorso, San Benedetto del Tronto, Ascoli Piceno
  - Ospedale generale regionale "F. Miulli", Acquaviva delle Fonti, Bari
  - Presidio Ospedaliero S. Maria delle Grazie, Pozzuoli, Napoli
  - AORN S.ANNA e S.SEBASTIANO, Caserta
  - Università degli Studi G. D'Annunzio, Chieti
  - Ospedale P. Monaldi, Napoli
  - Policlinico AO di Padova, Padua
  - Policlinico Universitario Campus Bio-Medico, Roma

DOCUMENTS (1):
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03489395/Prot_000.pdf